CLINICAL TRIAL: NCT05532449
Title: Low-dose Dezoxide Suppresses Sufentanil-induced Cough During Induction of General Anesthesia in Patients Undergoing Cardiac Surgery: a Prospective, Randomized, Controlled Trial
Brief Title: Dezoxide Suppresses Sufentanil-induced Cough
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022 Dezocine
Record Dates: First submitted 2022-09-01; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Sufentanil-induced Cough

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention)
- Dezocine (Experimental): intravenous dezocine (0.03mg/kg diluted to 5 ml)
  Interventions: Drug: Intravenous dizocine

INTERVENTIONS:
Drug: Intravenous dizocine — Intravenous dizocine (0.03mg/kg diluted to 5 ml)
  Arms: Dezocine

SUMMARY:
Dizocine (0.03 mg/kg) or saline followed by sufentanil 0.4ug/kg was administered, and induction was completed with 3 min of observation. Heart rate and mean arterial pressure (MAP) were recorded before induction of anesthesia, before and 1 min after intubation, and side effects during induction, such as vomiting, hypoxemia (SpO2 <90%), or other expected effects. The number of coughs was recorded in both groups, and the severity of cough was defined as follows: mild, 1-2 coughs; moderate, 3-4 coughs; severe, 5 or more coughs.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for elective valve surgery, artificial vessel replacement or coronary artery bypass graft surgery; Age 18~80 years old; Sex is not limited; ASA class II~III; NYHA Class II-III; Patients or their family members have signed the clinical trial informed consent form

Exclusion Criteria:

* Upper respiratory tract infection within the last two weeks; Long history of smoking; chronic obstructive pulmonary disease; Highly reactive airway diseases such as bronchitis and asthma; Presence of high cranial pressure, high eye pressure, pulmonary alveolus; Malignant tumor, hematological disease, severe liver and kidney dysfunction, recent serious infection, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2022-09-12 (Estimated); Primary Completion 2022-09-12 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
sufentanil-induced cough | 2 minutes after intubation
  rate and severity of cough after sufentanil injection

SECONDARY OUTCOMES:
heart rate | 2 minutes after intubation
  heart rate during induction of general anesthesia
mean arterial pressure | 2 minutes after intubation
  mean arterial pressure during induction of general anesthesia
SpO2 | 2 minutes after intubation
  SpO2 during induction of general anesthesia

IPD SHARING:
Plan to Share IPD: Undecided